CLINICAL TRIAL: NCT07164430
Title: The Impact of Infant and Maternal Immunoprophylaxis on Hospitalisation for Respiratory Syncytial Virus in the Australian Capital Territory: A Population-based Interrupted Time Series Study
Brief Title: The Impact of the 2025 Infant and Maternal Respiratory Syncytial Virus (RSV) Prevention Program on RSV-related Hospitalisations in the Australian Capital Territory
Status: Not yet recruiting | Type: Observational
Sponsor: Nicola Irwin (Other)
Responsible Party: Sponsor-Investigator, Nicola Irwin, Clinical Support Nurse, The Canberra Hospital
Organization: The Canberra Hospital (Other)
Other Study IDs: 2025.LRE.00223
Record Dates: First submitted 2025-09-04; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus (RSV) Infection; Respiratory Syncytial Virus Hospitalizations; Respiratory Syncytial Virus Immunization
Keywords: Interrupted Time Series Analysis; Epidemiologic Methods
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RSV cases: Children aged under 2 years with laboratory confirmed RSV infection

SUMMARY:
The goal of this observational study is to is to examine the impact of new RSV prevention medicines on the burden of RSV disease among young children. The main question it aims to answer is:

What was the impact of the 2025 RSV prevention program on RSV-related hospitalisation in children under 2 years of age?

Participants won't need to do anything additional for the study as only routinely collected health information will be used to answer the research question.

DETAILED DESCRIPTION:
Nirsevimab, a novel long-acting monoclonal antibody targeted at RSV became available for vulnerable babies in the Australian Capital Territory (a small jurisdiction in Australia) in April 2024. Maternal RSV vaccine, Abrysvo, became available for all women of 28-36 weeks gestation in February 2025. Through either nirsevimab or Abrysvo, all infants born from 1 January 2025 in the jurisdiction have universal eligibility for RSV immunoprophylaxis.

This study will use interrupted time series methodology to evaluate the impact of the 2025 RSV prevention program on RSV-related hospitalisation in children under 2 years of age. Historical data from 2022-2023 will form the pre-nirsevimab period, and 2022-2024 the pre-Abrysvo period. 2025 will form the post-intervention period.

Secondary objectives are to:

1. Evaluate the impact of the 2025 RSV prevention program on RSV-related Emergency Department (ED) presentations
2. Evaluate the impact on the reported incidence of RSV

ELIGIBILITY:
Inclusion Criteria:

* child aged under 2 years
* laboratory confirmed RSV

Exclusion Criteria:

* n/a

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study is set in the Australian Capital Territory, a small Australian jurisdiction with a single acute paediatric service provider.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
RSV Hospitalisation | At monthly time intervals over 3 years and 8 months
  RSV-related hospital admissions will be determined by reviewing hospital admissions occurring within one month of a positive RSV test. The discharge summary will be reviewed for a diagnosis or other clinical information consistent with RSV-related illness (bronchiolitis, respiratory tract infection, viral illness), and cross-checked with the ICD-10-AM coding for the episode.

SECONDARY OUTCOMES:
Emergency Department presentations | Monthly time intervals over a period of 3 years and 8 months
  RSV-related ED presentations will be determined by reviewing ED presentations occurring within one month of a positive RSV test. Documentation from the presentation will be reviewed for a discharge diagnosis or impression consistent with RSV-related illness (bronchiolitis, respiratory tract infection, viral illness). If no discharge letter or doctors' documentation is available, the triage note will be reviewed for a presenting complaint consistent with RSV-related illness (rhinorrhoea, nasal congestion, cough, respiratory distress, diffuse crackles and/or wheeze, fever, hypoxaemia, and associated feeding difficulties, vomiting, dehydration, or lethargy).
RSV cases | At monthly intervals over 3 years and 8 months
  RSV cases will be determined by laboratory notifications of positive RSV infection on PCR test to ACT Health, the body responsible for receiving notifiable disease notifications.

CONTACTS AND LOCATIONS:
Locations (1):
- The Canberra Hospital, Garran, Australian Capital Territory, Australia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD that underlie any published results may be shared upon reasonable request, and subject to ethics and governance processes.
Supporting Information: Study Protocol
Time Frame: From 3 months after publication of results to 3 years.
Access Criteria: Researchers with a methodologically sound proposal, subject to ethics and governance processes. A data sharing agreement will be required.
URL: https://www.act.gov.au/open/act-data-sharing-policy